CLINICAL TRIAL: NCT06488807
Title: Treatment of Perioperative Neurocognitive Disorders With Olfactory Enrichment: Study Protocol for a Randomized Controlled Trial
Brief Title: Treatment of Perioperative Neurocognitive Disorders With Olfactory Enrichment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Yuan Shen, MD, PhD, Director, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: dsyy008
Record Dates: First submitted 2024-06-15; First posted 2024-07-05 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Perioperative Neurocognitive Disorder
Keywords: Perioperative Neurocognitive Disorder; Odor Enrichment
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olfactory Enrichment Group (Experimental): All participants enrolled in the olfactory enrichment group will receive twice sessions per day with an interval of at least 6 hours on preoperative day 1 and postoperative day 1-3. Each session will last 30 minutes. Each participant will be equipped with an electrical odor dispenser which allowed to distribute 8 odors (grapefruit, lavender, lemon, peppermint, tangerine, green tea, cloves and eucalyptus). When pushing a button, 4 odors will be released in turn and participants will sniff each odor (approximately 4 ml odorized air) for approximately 30 seconds by a nasal catheter. Considering of the adaption of odors, 4 odors will be used in the morning session and another 4 odors will be used in the afternoon session.
  Interventions: Other: Olfactory Enrichment
- Sham Group (Sham Comparator): The sham group will receive sham olfactory enrichment sessions, which is designed with the same pattern (twice a day, 30 min for each session, on preoperative day 1 and on postoperative day 1-3. However, the containers provided to the sham group will be odorless. The odor containers and labels will appear identical to those used in the olfactory enrichment group.
  Interventions: Other: Sham

INTERVENTIONS:
Other: Olfactory Enrichment — Each participant will be equipped with an electrical odor dispenser which allowed to distribute 8 odors (grapefruit, lavender, lemon, peppermint, menthol, tangerine, green tea, and bergamot). The choice of odors was guided by (1) pleasantness of the odors, (2) presence of slight trigeminal activation in some of the odors, e.g., peppermint, (3) evaporation characteristics, so that the odors would last for the duration of the experiment, (4) technical issues mostly in terms of compatibility with the odor cartridge, (5) availability, and (6) inspiration from the previous studies.
  Arms: Olfactory Enrichment Group
Other: Sham — The containers provided to the sham group will be odorless. The odor containers and labels will appear identical to those used in the olfactory enrichment group.
  Arms: Sham Group

SUMMARY:
Perioperative neurocognitive disorder (PND) is one of the most common postoperative complications among elderly patients. However, the mechanism and targeted intervention of PND remains unclear. Our previous clinical studies demonstrated the association between olfactory impairment and PND. Moreover, our translational studies showed that anesthesia/surgery induced olfactory impairment and caused cognitive impairment in mice and olfactory enrichment could prevent the anesthesia/surgery-induced cognitive impairment. However, there was no clinical investigation to determine whether olfactory enrichment can mitigate PND in elderly patients. Therefore, we propose determining whether olfactory enrichment can prevent and/or treat PND in elderly patients.

DETAILED DESCRIPTION:
The study will be a double-blinded, randomized controlled trial. Participants (65 years old or older) undergoing scheduled orthopaedic surgery (≥2 hours, under general anesthesia) will be randomized to either olfactory enrichment group or sham group. Participants in olfactory enrichment group will receive olfactory enrichment with a dispenser twice sessions per day on preoperative day 1-3 and postoperative day 1-3 (30 min per session, 4 odors for each session) while participants in sham group will be equipped with the same pattern except that water will be used in the dispenser. Participants will be assessed twice daily by a research assistant blinded to allocation. The primary outcome will be the incidence of postoperative delirium measured by the Confusion Assessment Method on postoperative days 1, 2 and 3. The secondary outcomes will be the severity of postoperative delirium, cognitive function, plasma Tau-PT217 level, and olfactory function.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥65 years old.
2. Having a scheduled surgery (≥2 hours, general anesthesia) (e.g., total hip replacement, toal knee replacement, open reduction and internal fixation of hip and lumbar spine).
3. Being able to complete neuropsychological tests, 3D-CAM and CAM-S.
4. Chinese Mandarin as their native language.
5. Edmonton frailty scale (EFS) score ≥ 6.

Exclusion Criteria:

1. Having delirium, assessed by 3D-CAM, before surgery.
2. Having a brain tumour, stroke or mental disorders (eg, major depressive disorder or dementia).
3. Participating in other clinical studies at the time of screening.
4. Unwillingness to comply with the protocol or procedures.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 686 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | at baseline and postoperative day 1 to 3
  The presence of postoperative delirium will be defined according to 3D-CAM, which includes four entries: acute onset and fluctuating course, inattention, disorganized thinking and altered level of consciousness. To diagnose delirium, both the first and second criteria have to be present plus the third and/or fourth criteria. Every participant will be assessed twice daily after anesthesia/surgery from postoperative day 1 to postoperative day 3, with the first assessment between 8:00 and 10:00. The second assessment will be between 15:00 and 17:00.

SECONDARY OUTCOMES:
Incidence of delayed neurocognitive recovery and postoperative neurocognitive disorder | at baseline, on 21 days and 6 months after anesthesia/surgery
  Participants' cognitive function will be assessed at baseline, on postoperative day 21, and at postoperative month 6 using a battery of neuropsychological tests, including the Montreal Cognitive Assessment (MoCA), Hopkins Verbal Learning Test Retention (HVLTRet), Hopkins Verbal Learning Test Total Recall (HVLTTR), Brief Visuospatial Memory Test Total Recall (BVMTTR), Brief Visuospatial Memory Test Delayed Recall (BVMTDR), Benton Judgment of Line Orientation (JLO), Digit Span Test (DST), Verbal Fluency Test (VFT) and Trail Making Test (TMT). Cognitive Change Index will be calculated by subtracting baseline scores from postoperative scores in each of the neuropsychological tests. Delayed neurocognitive recovery or postoperative neurocognitive disorder will be defined as by a decrease by one or more standard deviations in at least two of the neuropsychological tests from the baseline to 21 days or 6 months after anesthesia/surgery.

OTHER OUTCOMES:
Severity of delirium | at baseline and postoperative day 1 to 3
  Severity of delirium will be assessed by the CAM-S. CAM-S includes 10 items: acute onset or symptom fluctuation, inattention, disorganized thinking, altered level of consciousness, disorientation, memory impairment, perceptual disturbances, psychomotor agitation, psychomotor retardation and sleep-wake cycle disturbance. Each item is scored as absent (0), mild (1) or marked (2), except acute onset or fluctuation, which is scored as absent (0) or present (1). The sum of CAM-S ranges from 0 (none) to 19 (most severe). The Delirium Symptom Interview (DSI) Daily will be used to determine CAM-S grades. The incidence of postoperative delirium will also be referred to the records by nurses on duty.
Severity of delayed neurocognitive recovery and postoperative neurocognitive disorder | at baseline, on 21 days and 6 months after anesthesia/surgery
  Severity of delayed neurocognitive recovery and postoperative neurocognitive disorder will be assessed by battery of neuropsychological tests at baseline, on postoperative day 21, and at postoperative month 6. The scores of neuropsychological tests indicate cognitive functions which can reflect the severity of delayed neurocognitive recovery and postoperative neurocognitive disorder.
Activities of Daily Living | at baseline, on 21 days and 6 months after anesthesia/surgery
  Activities of daily living will be assessed using the Chinese version of the ADL scale at baseline, and on postoperative day 21 days and 6 months after anesthesia/surgery, including a Physical Self-Maintenance Scale and an Instrumental Activities of daily living at baseline (before the surgery) and follow-ups. There are a total of 14 items in the Activities of daily living. For each item, scoring is determined by a 4-point coding system: 1 = 'can do it myself,' 2 = 'have some difficulty but can still do it by myself,' 3 = 'need help to do it,' and 4 = 'cannot do it at all.' A higher score therefore indicates greater impairment in activities of daily living. Specifically, a total activities of daily living score of 14 signifies no impairment, scores of 15-21 indicate mild impairment, and scores of ≥22 reflect severe impairment. Participants with Activities of daily living scores of more than 22 points will be considered to have substantive impairment in Activities of daily living.
Plasma Tau-PT217 Concentrations | immediately before and after anesthesia/surgery, 3 days, 21 days and 6 months postoperatively
  Five milliliters of blood will be collected from participants immediately before and after anesthesia/surgery, 3 days, 21 days and 6 months postoperatively. Blood samples will be centrifuged at 500 g for 10 minutes, and the plasma supernatant will be collected. The plasma will be collected in EDTA tubes, immediately placed on ice, and then stored in a -80°C freezer until analysis. The samples will be thawed at the time of measurement. Tau-PT217 concentrations in plasma will be measured using Nanoneedle technology.
Olfactory Function Determination | at baseline and on postoperative day 3, 21 and 6 months after anesthesia/surgery.
  Olfactory function will be assessed at baseline and on postoperative day 3, 21 and 6 months after anesthesia/surgery. The assessment will include odor threshold (scored from 1 to 20) and odor identification (scored from 0 to 16) tests, using pen-like odor dispensing devices to evaluate nasal chemosensory performance.

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Shen, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mei X, Wang J, Ni Z, Wang Y, Zhao B, Sessler DI, Xie Z, Shen Y. Effects of olfactory enrichment on perioperative neurocognitive disorders in elderly patients undergoing orthopedic surgery: a study protocol of a multi-center randomized controlled trial. Trials. 2025 Sep 26;26(1):363. doi: 10.1186/s13063-025-09109-w. PMID 41013688